CLINICAL TRIAL: NCT01456065
Title: A Phase I, Open, Randomized, Study to Investigate the Safety of Active Immunotherapy With Fully Mature, TERT-mRNA and Survivin - Peptide Double Loaded Dendritic Cells (DCs) in Subjects With Advanced Epithelial Ovarian Cancer, Enrolled in the Study Within Twelve Weeks After Completing Primary Therapy
Brief Title: Safety of Active Immunotherapy in Subjects With Ovarian Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Life Research Technologies GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LRT-I-L01 Ovar
Record Dates: First submitted 2011-09-14; First posted 2011-10-20 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine weekly administration (Other)
  Interventions: Biological: Procure
- Vaccine biweekly administration (Other)
  Interventions: Biological: Procure

INTERVENTIONS:
Biological: Procure — The IMP (Investigational Medical Product) consists of 1.3*107 autologous, fully mature DCs, double loaded with TERT-mRNA and Survivin-peptide, diluted in 0.5 mL of a standard freezing solution, made up of 10% DMSO (Dimethyl sulfoxide), solved in a physiologic water solution of 5% glucose; provided in a 2 mL cryovial. 8 vial will be injected on weekly administration basis to the patient.
  Arms: Vaccine weekly administration
Biological: Procure — The IMP consists of 1.3*107 autologous, fully mature DCs, double loaded with TERT-mRNA and Survivin-peptide, diluted in 0.5 mL of a standard freezing solution, made up of 10% DMSO, solved in a physiologic water solution of 5% glucose; provided in a 2 mL cryovial, 8 vials will be injected into the patient on biweekly basis.
  Arms: Vaccine biweekly administration

SUMMARY:
The purpose of this study is to investigate the safety of the active immune therapy based on the reiterated injection of fully mature, TERT (Telomerase Reverse Transcriptase)-mRNA and Survivin-peptide double loaded DCs (Dendritic Cells) [Procure®] in patients with advanced ovarian cancer, enrolled into the study within twelve weeks after completing primary therapy.

DETAILED DESCRIPTION:
This is an uncontrolled, randomized, parallel-group, open-label phase I trial in patients with advanced epithelial ovarian cancer. Patients were randomized into treatment group A with weekly administration versus treatment group B with bi-weekly administration.

Patients in both treatment groups received a maximum of eight injections administered one by one once a week for eight times for treatment group A and once in a fortnight for eight times for treatment group B.

The treatment was completed within seven weeks for Arm A and within 14 weeks for Arm B. Independently of the treatment arm they had been assigned to, all the patients were followed for a period covering a total of 12 or 19 weeks or until disease progression. Safety parameters (primary objective) and efficacy parameters (secondary objective) were recorded. Upon completion of the treatment, one follow-up visit took place at week 12 (group A, only) or 19 (group B, only).

To protect the patients' safety, the first six patients were treated as described below:

* The first patient was hospitalized and kept under medical observation for 72h after administration of the first and second dose of the investigational product;
* After an observational period of 3 days following the second dose of the first patient, the second and the third patient were administered the first dose of the investigational product, hospitalized and kept under medical observation for 72h. The two patients were treated simultaneously or consecutively;
* After an observational period of 3 days after the second dose to the first three patients, an interim safety report was sent to the Ethics Committee;
* Additionally the next three patients were hospitalized, administered their first dose of the vaccine and kept under medical observation for 72h. The three patients were treated simultaneously or consecutively.

  15 evaluable patients (which were randomized to one of the two treatment groups in equal numbers) 5 study sites in Austria and Hungary

ELIGIBILITY:
Inclusion criteria:

Patients with epithelial ovarian cancer FIGO (Fédération Internationale de Gynécologie et d'Obstétrique) stage III in remission after treatment with surgery (hysterectomy and ovariectomy) and after the first primary chemotherapy (standard treatment e.g. 6-9x Carboplatin/Taxane)

* Age > 18 ≤ 75 years
* Histological confirmed FIGO stage III ovarian epithelial cancer
* Stable disease at screening visit: negative CT and CA-125 within normal range
* Karnofsky status ≥ 70% and/or ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Life expectancy ≥ 6 months
* Adequate hematological function (WBC (white blood cells) ≥ 3000/µl, hemoglobin ≥ 10.0 g/dL, platelets > 100,000/µl)
* Adequate renal and hepatic function (serum creatinine ≤ 2.0 mg/dL, bilirubin total < 2 mg/dL, PT (INR) ≤ 1.5x institutional upper limit of normal)
* Signed and dated informed consent before the start of any study-specific procedure
* Body weight > 50 kg

Exclusion criteria:

* Surgery, radiation therapy or chemotherapy within eight weeks prior to leukapheresis
* Other biological therapy (Interferons, TNF (Tumor necrosis factors), Interleukins, mABs (Monoclonal antibodies), biological response modifiers) within eight weeks prior to undergo the leukapheresis
* History or presence of systemic autoimmune disease (such as, but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma or multiple sclerosis)
* Participation in other clinical trials or treatments with an investigational drug within four weeks prior to enrollment
* Serious intercurrent chronic or acute illness such as severe asthma or COPD (Chronic Obstructive Pulmonary Disease), cardiac (NYHA (New York Heart Association ) class III or IV) or hepatic disease, or other illness considered to constitute an unwarranted high risk for investigational drug treatment
* History of another malignancy within five years prior to study enrollment, except curatively treated non-melanotic skin cancer or cervical cancer in situ
* Presence of an active acute or chronic infection, including syphilis, HIV or viral hepatitis B and/or C
* Current treatment with corticosteroids (except of local) or other immunosuppressive agents such as azathioprine or cyclosporine A is excluded on the basis of its potential immune suppression. Any systemic steroid therapy must have been discontinued six weeks prior to undergo the leukapheresis
* Patients who have undergone organ transplantation
* Legally incapacitated persons and/or other circumstances, which make it difficult for the subject to understand the nature, meaning and consequences of the clinical study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events and clinical relevant deviations from Laboratory parameters | from first treatment until up to 12 to 19 weeks

SECONDARY OUTCOMES:
Number of circulating tumor cells in peripheral blood | from first treatment till up to 12 to 19 weeks
  Circulating tumor cells (CTCs) will be quantified prior vaccination and follow up. CTCs will be enriched from peripheral blood and characterized by specific biomarkers. Quantitation of CTCs will provide information about the stage of a malignancy, onset of disease progression and response of therapy.
Immune monitoring - Number of autologous dendritic cells loaded with tumor specific antigens | from first treatment until treatment visit 7 up to 12 weeks
  Immune monitoring will be done prior vaccination and during treatment. The immune reaction of the patients will be surveyed by determination of the frequency of specific markers for T-Cells, activated T-cells,B-cells,NK (Natural Killer)-cells, NKT (Natural Killer T)-cells.Quantification of these cells will be done by multicolour FACS (Florescence activated cell sorting). This method will be applied to determine the effects of dendritic cell treatment on the patients immune system.
time to progression (CA (Cancer Antigen)-125 and CT (Computer tomography) | from first treatment until up to 12 to 19 weeks
Overall survival | from first treatment until up to 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Imhof, Dr., Principal Investigator — Hospital Korneuburg
Locations (5):
- Austria (3):
  - Hospital Landeskrankenhaus Innsbruck, Innsbruck
  - Hospital Korneuburg, Korneuburg
  - Hospital Barmherzigen Schwestern, Linz
- Hungary (2):
  - Semelweis University, Budapest
  - National Oncology Institute, Budapest